CLINICAL TRIAL: NCT01729039
Title: Vestibular Rehabilitation and Dizziness in Geriatric Patients
Brief Title: Vestibular Rehabilitation and Dizziness
Acronym: DZO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E7613-R
Record Dates: First submitted 2012-11-13; First posted 2012-11-20 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Dizziness
Keywords: rehabilitation; aged; aged, 80 and over; vestibular diseases
MeSH Terms: conditions — Dizziness; Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- gaze stability (Experimental): standard balance rehabilitation plus vestibular-specific exercises
  Interventions: Behavioral: standard balance rehabilitation; Behavioral: gaze stability
- control (Placebo Comparator): standard balance rehabilitation plus placebo eye exercises
  Interventions: Behavioral: standard balance rehabilitation; Behavioral: Control

INTERVENTIONS:
Behavioral: standard balance rehabilitation — All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility with progressively challenging tasks. Balance exercises include maintaining stability with vision and somatosensory cues altered, dynamic weight shifts and performing ankle, hip and step strategies. Gait activities include negotiating uneven terrains and obstacles, gait with head turns, varied speed, and unpredictable starts and stops. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
Behavioral: gaze stability — Vestibular adaptation and substitution exercises will be performed by the experimental group (GS). Adaptation exercises involve head movement while maintaining focus on a target, which may be stationary or moving. Typical progression of adaptation exercises involve increased velocity of head movement, movement of both target and head, target placed in a distracting visual pattern and maintenance of a challenging posture. During active eye-head exercise, a large eye movement to a target is made prior to the head moving to face the target, potentially facilitating use of preprogrammed eye movements.
  Arms: gaze stability
Behavioral: Control — The placebo exercises will consist of saccadic eye movements while the head is stationary and will be performed by the control group. These eye movements will be performed against a plain background in order to eliminate retinal slip and, therefore, eliminate the error signal for vestibular adaptation.
  Arms: control

SUMMARY:
The purpose of this study is to determine whether vestibular exercises provide added benefit to balance rehabilitation in older adults with dizziness and normal vestibular function.

DETAILED DESCRIPTION:
Dizziness is among the most prevalent complaints for which people seek medical help and the incidence increases with advancing age. Dizziness represents a diagnostic and treatment challenge because it is a subjective sensation, refers to a variety of symptoms (unsteadiness, spinning, sense of motion or lightheadedness), and has many potential contributory factors. Dizziness is often related to vestibular disease which is treated effectively with vestibular exercises. Successful management of dizziness is critical because dizziness is a major risk factor for falls in older adults.

There are parallels between the effects of age-related versus disease-related loss of vestibular function - in complaints of dizziness and increased risk for falls. The investigators' question, then, is whether the same exercises that are beneficial for patients with vestibular pathology are beneficial for older patients with dizziness but normal vestibular function.

Older adults with dizziness who have been referred to Audiology for vestibular evaluation will be randomized to receive either standard balance rehabilitation plus placebo eye exercises (CON) or standard balance rehabilitation plus vestibular-specific exercises (GS). Primary outcomes include symptoms, balance-related confidence, dynamic visual acuity, postural stability as measured by sensory organization test, fall risk as measured by dynamic gait index, and gait speed. Assessment will occur at baseline, discharge from physical therapy (PT), 1 and 6 months post-PT.

ELIGIBILITY:
Inclusion Criteria:

* at least 50 years of age
* documented balance or mobility problems
* normal vestibular function, including otolith function

Exclusion Criteria:

* cognitive impairment
* progressive medical issues that would impact mobility (e.g., Parkinson's disease, cerebellar atrophy)
* dizziness due to orthostatic hypotension or Benign Paroxysmal Positional Vertigo (BPPV)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Hall, PhD PT, Principal Investigator — Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN
Locations (2):
- United States (2):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Mountain Home VA Medical Center James H. Quillen VA Medical Center, Mountain Home, TN, Mountain Home, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Gaze Stability: Standard balance rehabilitation plus Vestibular-specific exercises
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Vestibular-specific exercises: Gaze stability exercises are performed by the experimental group (GS). Adaptation exercises involve head movement while maintaining focus on a target. Progression involves increased velocity of head movement and target placed in a distracting visual pattern and maintenance of a challenging posture. During active eye-head exercise, a large eye movement to a target is made prior to the head moving to face the target.
- Control: Standard balance rehabilitation plus Placebo eye exercises
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Control: Placebo exercises consist of saccadic eye movements while the head is stationary and are performed by the control group (CON). These eye movements are performed against a plain background in order to eliminate retinal slip and, therefore, eliminate the error signal for vestibular adaptation.
Period: Overall Study
Arm/Group | Gaze Stability | Control
Started | 23 | 26
Completed | 13 | 14
Not Completed | 10 | 12
Not completed — disqualified | 2 | 5
Not completed — Withdrawal by Subject | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Gaze Stability (GS): Gaze Stability group intervention includes standard balance rehabilitation plus vestibular-specific exercises.
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Vestibular-specific exercises: Gaze stability exercises involve head movement while maintaining focus on a target. Progression involves increased velocity of head movement and target placed in a distracting visual pattern and maintenance of a challenging posture. During active eye-head exercise, a large eye movement to a target is made prior to the head moving to face the target.
- Control (CON): Control group intervention includes standard balance rehabilitation plus placebo eye exercises.
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Control exercises: Placebo eye exercises consist of saccadic eye movements while the head is stationary. These eye movements are performed against a plain background in order to eliminate retinal slip and, therefore, eliminate the error signal for vestibular adaptation.
- Total: Total of all reporting groups
Arm/Group | Gaze Stability (GS) | Control (CON) | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.85 (8.80) | 72.36 (6.07) | 71.15 (7.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Visual Analog Scale - Head Movement [Mean (Standard Deviation); unit: units on a scale] — This scale was used to measure perceived level of dizziness after one minute of horizontal head movement at 1 Hz. This technique uses a 10-cm line with one end being no symptoms (score = 0) and the other representing the worse possible symptoms (score = 10) and is commonly used to assess perception of pain. The subject is asked to place a mark on the 10-cm line at a point which indicates the intensity of his/her perception of symptoms of dizziness and the distance along that line is measured. Scores range from 0 to 10 with higher scores indicating worse perceived dizziness.
  units on a scale | 2.06 (2.69) | 2.58 (2.74) | 2.33 (2.68)
Visual Analog Scale - Disequilibrium [Mean (Standard Deviation); unit: units on a scale] — This scale was used to measure perceived level of unsteadiness while walking. This technique uses a 10-cm line with one end being no symptoms (score = 0) and the other representing the worse possible symptoms (score = 10) and is commonly used to assess perception of pain. The subject is asked to place a mark on the 10-cm line at a point which indicates the intensity of his/her perception of symptoms of unsteadiness and the distance along that line is measured. Scores range from 0 to 10 with higher scores indicating worse perceived unsteadiness.
  units on a scale | 1.77 (1.69) | 2.74 (2.10) | 2.29 (1.95)
Dynamic Gait Index [Mean (Standard Deviation); unit: units on a scale] — The dynamic gait index (DGI) assesses an individual's ability to modify balance while walking in the presence of external demands. The 8 items of the DGI include walking while changing speed and turning the head, walking over and around obstacles, and stair climbing. Scoring of the DGI is based on a 4-point scale from 0 to 3 with 0 indicating severe impairment and 3 indicating normal ability. A maximum total score of 24 is possible and scores of < 20 indicate high risk for falling.
  units on a scale | 18.46 (3.15) | 18.36 (2.62) | 18.41 (2.83)
Activities-specific balance confidence scale [Mean (Standard Deviation); unit: percentage] — As a result of their disequilibrium, subjects report decreased confidence that they can maintain their balance in a variety of situations. The Activities-specific balance confidence scale (ABC) was developed to measure confidence with balance across a range of 16 activities of increasing challenge. Items are rated on a rating scale that ranges from 0 - 100% with a score of zero representing no confidence and a score of 100 representing complete confidence. An overall score is calculated by averaging the items with higher scores indicating higher (better) balance confidence.
  percentage | 69.64 (21.12) | 78.03 (9.68) | 74.00 (16.42)
10 Meter Walk Test [Mean (Standard Deviation); unit: ft/s] — This measure assesses walking speed over a short distance. Subjects were asked to walk at their preferred gait speed for a distance of 30 feet which allowed 5 feet for acceleration and deceleration at the beginning and end of the walk. The time it took to walk 20 feet was recorded using a calibrated stopwatch and gait speed (ft/s) was calculated.
  ft/s | 3.05 (0.58) | 2.96 (0.58) | 3.00 (0.57)

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale - Head Movement
Description: This scale was used to measure perceived level of dizziness after one minute of horizontal head movement at 1 hertz (Hz). This technique uses a 10-cm line with one end being no symptoms (score = 0) and the other representing the worse possible symptoms (score = 10) and is commonly used to assess perception of pain. The subject is asked to place a mark on the 10-cm line at a point which indicates the intensity of his/her perception of symptoms of dizziness and the distance along that line is measured. Scores range from 0 to 10 with higher scores indicating worse perceived dizziness.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Gaze Stability: Gaze stability (GS) group intervention includes standard balance rehabilitation plus vestibular-specific exercises
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Vestibular-specific exercises: Gaze stability exercises include adaptation exercises which involve head movement while maintaining focus on a target. Typical progression involves increased velocity of head movement and target placed in a distracting visual pattern. During active eye-head exercise, a large eye movement to a target is made prior to the head moving to face the target.
- Control: Control group (CON) intervention includes standard balance rehabilitation plus placebo eye exercises.
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Placebo eye exercises: Saccadic eye movements are performed while the head is stationary. These eye movements are performed against a plain background in order to eliminate retinal slip and, therefore, eliminate the error signal for vestibular adaptation.
Arm/Group | Gaze Stability | Control
Number analyzed (Participants) | 13 | 14
units on a scale | 1.56 (2.55) | 1.81 (2.08)
Statistical Analysis 1: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .356, ANOVA — Main effect of time (baseline to post-PT) alpha = .05
Statistical Analysis 2: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .840, ANOVA — Interaction of Time by Group (GS vs. CON) alpha = .05

2. Primary Outcome: Visual Analog Scale - Disequilibrium
Description: This scale was used to measure perceived level of unsteadiness while walking. This technique uses a 10-cm line with one end being no symptoms (score = 0) and the other representing the worse possible symptoms (score = 10) and is commonly used to assess perception of pain. The subject is asked to place a mark on the 10-cm line at a point which indicates the intensity of his/her perception of symptoms of unsteadiness and the distance along that line is measured. Scores range from 0 to 10 with higher scores indicating worse perceived unsteadiness.
Time Frame: 6 weeks
Population: Repeated Measure (RM) ANOVA
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gaze Stability | Control
Number analyzed (Participants) | 13 | 14
units on a scale | 1.66 (2.29) | 1.96 (2.37)
Statistical Analysis 1: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .170, ANOVA — Main effect of Time (baseline to post-PT) Alpha=.05
Statistical Analysis 2: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .297, ANOVA — Interaction of Time by Group (GS vs. CON) alpha = .05

3. Secondary Outcome: Dynamic Gait Index
Description: The dynamic gait index (DGI) assesses an individual's ability to modify balance while walking in the presence of external demands. The 8 items of the DGI include walking while changing speed and turning the head, walking over and around obstacles, and stair climbing. Scoring of the DGI is based on a 4-point scale from 0 to 3 with 0 indicating severe impairment and 3 indicating normal ability. A maximum total score of 24 is possible and scores of < 20 indicate high risk for falling.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Control: Control (CON) group intervention includes standard balance rehabilitation plus placebo eye exercises.
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Placebo eye exercises: Saccadic eye movements are performed while the head is stationary. These eye movements are performed against a plain background in order to eliminate retinal slip and, therefore, eliminate the error signal for vestibular adaptation.
Arm/Group | Gaze Stability | Control
Number analyzed (Participants) | 13 | 14
units on a scale | 21.54 (2.02) | 21.21 (2.78)
Statistical Analysis 1: Comparison: Gaze Stability vs Control; Test type: Superiority; p < .001, ANOVA; Main effect of Time (baseline to post-PT) alpha = .05
Statistical Analysis 2: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .817, ANOVA — Interaction of Time by Group (GS vs. CON) alpha = .05

4. Secondary Outcome: Activities-specific Balance Confidence Scale
Description: As a result of their disequilibrium, subjects report decreased confidence that they can maintain their balance in a variety of situations. The Activities-specific balance confidence scale (ABC) was developed to measure the subject's confidence with their balance across a range of 16 activities of increasing challenge. Items are rated on a rating scale that ranges from 0 - 100% with a score of zero representing no confidence and a score of 100 representing complete confidence. An overall score is calculated by averaging the items with higher scores indicating higher (better) balance confidence.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Gaze Stability | Control
Number analyzed (Participants) | 13 | 14
percentage | 83.98 (14.40) | 83.37 (6.30)
Statistical Analysis 1: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .005, ANOVA — Main effect of Time (baseline to post-PT) alpha = .05
Statistical Analysis 2: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .172, ANOVA — Interaction of Time by Group (GS vs. CON) alpha = .05

5. Secondary Outcome: 10 Meter Walk Test
Description: This measure assesses walking speed over a short distance. Subjects were asked to walk at their preferred gait speed for a distance of 30 feet which allowed 5 feet for acceleration and deceleration at the beginning and end of the walk. The time it took to walk 20 feet was recorded using a calibrated stopwatch and gait speed (ft/s) was calculated.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: ft/s
Arm/Group | Gaze Stability | Control
Number analyzed (Participants) | 13 | 14
ft/s | 3.15 (0.54) | 3.28 (0.69)
Statistical Analysis 1: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .009, ANOVA — Main effect of time (baseline to post-PT) alpha = .05
Statistical Analysis 2: Comparison: Gaze Stability vs Control; Test type: Superiority; p = .146, ANOVA — Interaction of Time by Grou (GS vs. CON) alpha = .05

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Control: Control group (CON intervention includes standard balance rehabilitation plus placebo eye exercises.
  Standard balance rehabilitation: All subjects perform balance and gait exercises in addition to eye exercises and receive a written home exercise program (HEP) of balance and gait exercises to improve postural stability and mobility. Walking for endurance is included in the HEP. Each participant receives a customized balance and gait HEP based on identified impairments and is progressed according to ability and level of assistance at home.
  Placebo eye exercises: Saccadic eye movements are performed while the head is stationary. These eye movements are performed against a plain background in order to eliminate retinal slip and, therefore, eliminate the error signal for vestibular adaptation.
Arm/Group | Gaze Stability | Control
All-Cause Mortality (participants affected / at risk) | 1/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gaze Stability (N=23) | Control (N=26)
Fall resulting in fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Fall while performing home exercise program
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gaze Stability (N=23) | Control (N=26)
Fall without injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Loss of balance without injury while performing home exercise program

LIMITATIONS AND CAVEATS:
High dropout rate; small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes